CLINICAL TRIAL: NCT01649050
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Parallel-group Study to Assess the Efficacy of 5 Weeks of Treatment With BGG492 in Patients With Spasticity Due to Multiple Sclerosis
Brief Title: Efficacy of 5 Weeks of Treatment With BGG492 in Patients With Spasticity Due to Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBGG492A2215; 2012-002783-27 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-07-25 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2014-08

CONDITIONS: Muscle Spasticity Due to Multiple Sclerosis
Keywords: Spasticity; Multiple Sclerosis
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis | interventions — selurampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BGG492 (Experimental): BGG492 tablets administered orally
  Interventions: Drug: BGG492
- Placebo (Placebo Comparator): Matching placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGG492
  Arms: BGG492
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate efficacy and safety of BGG492 versus placebo on moderate to severe spasticity due to multiple sclerosis

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of multiple sclerosis (MS) of any type.
* MS diagnosis at least 6 months prior to screening.
* Stable MS with no relapse within 3 months prior to screening.
* Treated or untreated spasticity due to MS for at least 3 months prior to screening, not wholly relieved with antispasticity medications.

Key exclusion criteria:

* Patients with symptoms of spasticity not due to MS.
* Patients taking three or more different anti-spasticity medications.
* Acute MS exacerbation requiring treatment within 3 months of the Screening Visit.
* Initiation of, or the discontinuation of interferon beta or any other disease modifying therapy for MS within 3 months of the Screening Visit.
* Use of baclofen pump at any time.
* Wheelchair or bed-bound patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in spasticity NRS score from baseline to 5 weeks | 5 weeks
  The spasticity Numeric Rating Scale is a 0 to 10 patient reported scale of spasticity severity, with 0 being no spasticity and 10 being worst possible spasticity.
PGIC score at 5 weeks | 5 weeks
  The Patient Global Impression of Change is a patient reported one item mesaure of overall improvement in condition since the previous visit. The patient is asked to choose one of 7 sentences from very much improved to very much worse, that best describes his present condition.

SECONDARY OUTCOMES:
Change from baseline to 5 weeks in Ashworth spasticity score | 5 weeks
  The Ashworth spasticity score is a physician assessed rating of spasticity using a five point score from 0 to 4 for each muscle group tested.
Safety and tolerability | average of 70 days, maximum from day -19 to day 52, i.e. from first baseline up to study completion visit
  Number of patients with adverse events (AE).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals